CLINICAL TRIAL: NCT06732375
Title: Pilot Study of Mindset Moments Among Adolescent and Young Adult Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00116490
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Youth Cancer; Young Adult Cancer; Distress, Psychological
Keywords: young adult cancer survivor; distress; youth cancer survivor; resilience
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): Study participation will involve attending 8 weekly, one hour, live online group sessions and completing daily 5 minute activities such as guided imageries and CBT (cognitive behavioral therapy) check-in within the app.
  Interventions: Behavioral: Mindset Moments

INTERVENTIONS:
Behavioral: Mindset Moments — MM™ includes: 1) CBT; 2) resilience training; 3) mindfulness-based stress reduction; 4) peer support; and 5) family conversations delivered in small virtual groups, with a "mentor" who facilitates resilience-building conversations prompted from "Skill of the Week" lessons.

SUMMARY:
The purpose of this study is to evaluate the feasibility and acceptability of the Mindset Moments™ (MM™) program in managing psychological distress and resiliency in adolescent and young adult cancer survivors.

Study participation will involve attending 8 weekly, one hour, live online group sessions and completing daily 5 minute activities such as guided imageries and CBT check in within the app. Participants will also be asked to complete an online survey at the time of enrollment and at 4 and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 19-25 years of age
* Prior AYA cancer diagnosis
* Completed primary treatment for their cancer
* Score of 3 or above on the Distress Thermometer at the time of recruitment

Exclusion Criteria:

* Individuals without legal capacity to give consent
* Individuals who are not fluent in reading, writing, and speaking English

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Anxiety as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) | 8 weeks
  8-measure short form to assess the severity of anxiety symptoms within the Patient-Reported Outcomes Measurement Information System (PROMIS) framework. The total score ranges from 8 to 40, where a higher score indicates greater anxiety.

SECONDARY OUTCOMES:
Depression as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) | 8 weeks
  8-measure short form to assess the severity of anxiety symptoms within the Patient-Reported Outcomes Measurement Information System (PROMIS) framework. The total score ranges from 8 to 40, where a higher score indicates greater depression.
Symptoms of Post-Traumatic Stress Disorder (PTSD) as measured by the PCL-5 | 8 weeks
  The PTSD Checklist for DSM-V (PCL-5) is a self-report measure that assesses symptoms of PTSD. The total score ranges from 0 to 80, where a higher score indicates a greater severity of PTSD symptoms
Distress as measured by the National Comprehensive Cancer Network's (NCCN) Distress Thermometer (DT) | 8 weeks
  The NCCN DT is a tool that helps identify and address distress in cancer patients. The DT is a self-reported, 11-point scale that measures distress over the past week. The scale ranges from 0 (no distress) to 10 (extreme distress).
Ability to deal with stressful situations as measured by the Shift-and-Persist Scale | 8 weeks
  The Shift-and-Persist Scale has 14 items that measure two strategies for dealing with stressful situations: shifting, which means accepting stress and getting used to it; and persisting, which means being optimistic and finding purpose in tough times. The total score ranges from 8 to 32, where a higher score indicates a greater ability to deal with stressful situations.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia K Smith, PhD, MSW, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No